CLINICAL TRIAL: NCT01773018
Title: A Phase I, Open-label, Dose-escalation Study of the Safety and Pharmacokinetics of HMPL-504 in Patients With Advanced Solid Tumors
Brief Title: Phase I Study of the Volitinib (HMPL-504) in Patients With Advanced Solid Tumors
Acronym: HMPL-504
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hutchison Medipharma Limited (Industry)
Collaborators: Sir Charles Gairdner Hospital (Other); Austin Hospital, Melbourne Australia (Other); Monash University (Other)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-504-00AU1
Record Dates: First submitted 2013-01-15; First posted 2013-01-21 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Tumor
MeSH Terms: conditions — Neoplasms | interventions — 1-(1-(imidazo(1,2-a)pyridin-6-yl)ethyl)-6-(1-methyl-1H-pyrazol-4-yl)-1H-(1,2,3)triazolo(4,5-b)pyrazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Volitinib(HMPL-504) (Experimental): There are six dose cohorts,including 100, 200, 400, 600,800 and 1000 mg/day, HMPL-504 will be administered orally to patients once daily for each dose cohort.
  An alternative dosing schedule of twice every day (BID) may be investigated if pharmacokinetic studies indicate faster than anticipated clearance of Volitinib(HMPL-504).
  Interventions: Drug: Volitinib

INTERVENTIONS:
Drug: Volitinib — Volitinib(HMPL-504) is a tablet in the form of 25 mg ,100mgand 200 mg,oral,once daily.
  Other Names: HMPL-504

SUMMARY:
Volitinib (HMPL-504) is a novel, highly potent and selective small molecule inhibitor of c-Met kinase. In preclinical studies, it demonstrated strong in vitro and in vivo activity against c-Met kinase and its downstream signaling targets and inhibited tumor cell growth. This first-in-human study is conducted to assess the maximum tolerated dose (MTD) and dose-limiting toxicity (DLT), to evaluate the pharmacokinetics, safety and preliminary anti-tumor activity of HMPL-504 at single doses and multiple doses.

DETAILED DESCRIPTION:
This is a Phase I, first-in-human, open-label, dose-escalation study of Volitinib (HMPL-504) administered orally once every day(QD) to patients with locally advanced or metastatic solid tumors.There are two stages to this study : a dose-escalation stage and a dose-expansion stage. The dose-escalation stage is designed to evaluate the safety, tolerability, and pharmacokinetics of single dose and repeat doses of HMPL-504 given once every day (QD). An alternative dosing schedule of twice every day (BID) may be investigated if pharmacokinetic studies indicate faster than anticipated clearance of HMPL-504.

All patients will be carefully followed for adverse events during the study treatment and for 30 days after the last dose of study drug. Subjects of this study will be permitted to continue therapy with only safety monitoring and bimonthly assessments for progression, if the product is well tolerated and the subject has stable disease or better.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Age≥18 years
* Histologically or cytologically documented, incurable, locally advanced, or metastatic solid malignancy that has progressed on, or failed to respond to, at least one prior systemic therapy
* Evaluable or measurable disease per Response Evaluation Criteria in Solid Tumors(RECIST)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, or 1
* Male or female patients of child-producing potential must agree to use double barrier contraception, condoms, sponge, foams, jellies, diaphragm or intrauterine device (IUD), contraceptives (oral or parenteral), Implanon, injectables or other avoidance of pregnancy measures during the study and for 90 days after the last day of treatment
* In the dose expansion stage, the patient's informed consent to providing fresh biopsy tumor sample at baseline and day 7 should be obtained. Patients with gastric cancer , NSCLC, colorectal cancer, breast cancer and hepatocellular carcinoma(HCC) are preferred to be enrolled into the dose expansion cohort.

Exclusion Criteria:

• Inadequate hematologic and organ function, defined by the following (hematologic parameters must be assessed ≥14 days after a prior treatment, if any):

* Absolute neutrophil count <1500 cells/L
* Hemoglobin <9 g/dL
* Total bilirubin >1.5 × the upper limit of normal （ULN） with the following exception: Patients with known Gilbert disease who have

serum bilirubin level ≤3× the upper limit of normal（ULN） and normal AST/ALT may be enrolled.

* Aspartate aminotransferase （AST） and/or Alanine transaminase（ALT） >2.5 × the upper limit of normal（ULN） with the following exception: Patients with documented liver metastases may have AST and/or ALT levels ≤5 ×the upper limit of normal（ULN）.
* Serum creatinine >1.5 × the upper limit of normal (ULN) with the following exception: A creatinine clearance of ≥50 mL/min based on a documented 24-hour urine collection.
* International normalized ratio (INR)>1.5× the ULN or activated partial thromboplastin time (aPTT)>1.5×the ULN
* The INR applies only to patients who do not receive therapeutic anti-coagulation.

  • Any anti-cancer therapy, including chemotherapy, hormonal therapy, biologic therapy, radiotherapy, or herbal therapy within 4 weeks prior to initiation of study treatment with the following exceptions:
* Hormonal therapy with gonadotropin-releasing hormone (GnRH) agonists for prostate cancer
* Hormone-replacement therapy or oral contraceptives
* Palliative radiation to bone metastases > 2 weeks prior to Day 1
* Herbal therapy >1 week prior to Day 1

  * Adverse events from prior anti-cancer therapy that have not resolved to Grade ≤ 1, except for alopecia
  * Clinical significant active infection
  * Known clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis
  * Known human immunodeficiency virus infection
  * Pregnant (positive pregnancy test) or lactating women
  * New York Heart Association (NYHA) Class II or greater congestive heart failure
  * History of myocardial infarction or unstable angina within 6 months prior to Day 1
  * History of stroke or transient ischemic attack within 6 months prior to Day 1
  * Active or untreated brain metastasis
  * Inability to take oral medication, prior surgical procedures affecting absorption, or active peptic ulcer disease
  * Inability to comply with study and follow-up procedures
  * Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding that, in the investigator's opinion, gives reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or renders the patient at high risk from treatment complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2012-02; Primary Completion 2015-12 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
The safety and tolerability of single and multiple doses of HMPL-504 administered to patients. | up to 20 months
  The primary endpoint is evaluation of safety and tolerability during all the study of therapy following the initiation of multiple dosing of HMPL-504. The safety and tolerability variables to be evaluated in this study are adverse events, physical examinations, vital signs (specifically including blood pressure), clinical laboratory evaluations including serum chemistry, hematology(Maximum Tolerated Dose) , and urinalysis (with detailed sediment analysis, proteinuria, and 24-hour urine for collection for protein), and electrocardiograms (ECGs) in triplicate,Incidence and nature of DLTs(Dose-Limiting Toxicity),To determine the MTD (Maximum Tolerated Dose).

SECONDARY OUTCOMES:
Pharmacokinetic Assessments for area under curve (AUC), Cmax and Tmax . | Day 1-3 Single Dose and Day 1-21 Steady State
  In the study of single-dose, full Pharmacokinetics(PK) profiles of HMPL-504 will be obtained following administration of a single oral dose of HMPL-504 on Day 1 to Day 3. At multiple-dose, Pharmacokinetics(PK) sampling will include a pre-dose and at the 0.5,2,4,6,8 hour time points on days 1,15,21of dosing in the first 21-Day cycle of therapy, and pre-dose on days 2,8,16,and 22 of the first 21-Day cycle of therapy

OTHER OUTCOMES:
Objective Response Rate （ORR) | participants will be followed for the duration of hospital stay,an expected average of 3 months.
  Anti-tumoral efficacy will be assessed by best radiographic response based on Response Evaluation Criteria in Solid Tumors at baseline (Day -14 to -1) and at the end of two 21-Day cycles of therapy . For patients that continue on repeat 21-Day cycles after the primary evaluation period, progression will be assessed after each one 21-Day cycles of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Michael Millward, MD,Ph.D, Principal Investigator — Sir Charles Gairdner Hospital & University of WA; Hui Gan, MD,Ph.D, Principal Investigator — Austin Hospital, Melbourne Australia; Jason Lickliter, MD,Ph.D, Principal Investigator — Southern Health and Monash Institute of Medical Research
Locations (3):
- Australia (3):
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - Southern Health and Monash Institute of Medical Research, Clayton
  - Austin Health, Melbourne

IPD SHARING:
Plan to Share IPD: No